CLINICAL TRIAL: NCT01897740
Title: A LOCAL, SINGLE-CENTRE, EXTENSION, OPEN LABEL ACCESS STUDY, TO PROVIDE SILDENAFIL THERAPY FOR SUBJECTS WHO COMPLETED A1481156 STUDY AND ARE JUDGED BY THE INVESTIGATOR TO DERIVE CLINICAL BENEFIT FROM CONTINUED TREATMENT WITH SILDENAFIL, PRIOR TO REIMBURSEMENT AND AVAILABILITY FOR SUBJECTS IN RUSSIAN FEDERATION
Brief Title: Sildenafil Therapy For Subjects Who Derive Clinical Benefit From Continued Treatment With Sildenafil
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1481307
Record Dates: First submitted 2013-07-08; First posted 2013-07-12 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: sildenafil; pulmonary arterial hypertension; PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Sildenafil Citrate

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: sildenafil — tablets of sildenafil 20 mg 3 times a day for subjects with body weight > 20 kg and 10 mg TID for subjects with body weight ≤ 20 kg. If subject is 18 years of age or older, the recommended dose is 20 mg TID, regardless of body weight.

SUMMARY:
The purpose of this study is to provide Sildenafil therapy for subjects who completed A1481156 study and are judged by the investigator to derive clinical benefit from continued treatment with Sildenafil, prior to reimbursement and availability for subjects in the Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* Patients Who Completed study A1481156 and Are Judged by the Investigator to Derive Clinical Benefit from Continued Treatment with Sildenafil, Prior to Reimbursement and Availability for Subjects in Russian Federation.
* Child bearing age women should have appropriate contraception.
* Signed informed consent. Patients who have a wish and possibility to follow treatment regimens in terms of the study.

Exclusion Criteria:

* Pregnant and lactating women.
* Participation in other studies in the current moment or during study period except of A1481156.
* Patients with severe acute or chronic diseases psychiatric disorders or laboratory abnormalities.

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Moscow Research Institute of Pediatrics and Pediatric Surgery, Moscow, Russia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481307&StudyName=Sildenafil%20Therapy%20For%20Subjects%20Who%20Derive%20Clinical%20Benefit%20from%20Continued%20Treatment%20With%20Sildenafil